CLINICAL TRIAL: NCT04494763
Title: Propanolol for Primary Prophylaxis for Variceal Bleed in Biliary Atresia - An Open Label Randomized Controlled Study
Brief Title: Primary Prophylaxis for Variceal Bleed in Biliary Atresia
Acronym: BA-BB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ILBS-PHT-BA01
Record Dates: First submitted 2018-04-19; First posted 2020-07-31 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2020-07

CONDITIONS: Portal Hypertension, Biliary Atresia
Keywords: Variceal bleed; primary prophylaxis; Biliary atresia
MeSH Terms: conditions — Hypertension, Portal; Biliary Atresia | interventions — Propranolol

STUDY DESIGN:
Intervention Model Description: Open label Randomized controlled trial - Block randomization
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Propanolol (Experimental): Dose: 1 to 8 mg/kg/day in 1 to 2 divided doses adjusted to achieve target reduction in resting heart rate by 25% from baseline Frequency: once to Twice daily Route of Administration: Oral Duration: 18 months
  Interventions: Drug: Propanolol
- Placebo (Placebo Comparator): Placebo in a similar manner
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Propanolol — Non-selective Beta-blocker
  Arms: Propanolol
Other: Placebo — Inactive drug
  Arms: Placebo

SUMMARY:
Biliary atresia is the commonest etiology of neonatal cholestasis and is the most common indication for pediatric liver transplantation world-wide. Kasai-portoenterostomy (KPE) is the operative procedure of choice which helps in restoration of biliary flow and preventing rapid progression of fibrosis. Only 50-60% of infants have a successful surgery in terms of normalization of bilirubin (<2 mg/dL) after 3 months. Remaining 40-50% have rapid progression of PHT and eventual decompensation. Additionally, around 50-70% of infants with successful KPE have 1 or more episodes of cholangitis, and the severe ones if left untreated lead to progressive portal hypertension. Moreover in Indian setting a significant number of infants with biliary atresia reach late when the KPE is not feasible, and this group develops very rapid PHT and decompensation. Hence, overall around 70-80% of infants and children develop PHT within 5 years of age. Variceal bleed has been shown to be an important determinant of survival in infants with high bilirubin. Usage of beta-blockers in adult cirrhotics has been shown to reduce the progression of varices and incidence of variceal bleed. Although many pediatric hepatology centers worldwide use beta-blockers, there has been no controlled trial specifically to address this issue in children with biliary atresia. So, we planned this study to evaluate the efficacy of beta-blockers as primary prophylaxis for prevention of variceal bleed in biliary atresia children.

DETAILED DESCRIPTION:
(a) Aim and Objectives:

Aim: To study the effect of beta-blockers for primary prophylaxis of variceal bleed in infants and children with biliary atresia.

Primary objective: Bleeding free survival over 18 months FU

Secondary objectives:

(i) Progression, persistence or regression of esophageal and gastric varices, and portal hypertensive gastropathy over 3, 6, 12 and 18 months FU

(ii) Overall survival at 18 months FU

(b) Methodology: This will be an open label randomized controlled study where infants and children with biliary atresia from 6 months to 5 years fulfilling inclusion and exclusion criteria will be enrolled to receive propanolol or placebo for a duration of 18 months or till the occurrence of variceal bleed.

i. Study design: Open label randomized controlled study with stratified randomization.

ii. Intervention: Beta-blocker (Propanolol) versus placebo.

iii. Study period: 1.5 years

iv. Study population: Infants and children from 6 months to 5 years of age with Biliary atresia fulfilling the inclusion and exclusion criteria.

(c) Expected outcome of the project: Beta-blockers reduce the incidence of variceal bleed in infants and children with biliary atresia.

ELIGIBILITY:
Inclusion Criteria: Infants and children with biliary atresia from 6 months to 5 years of age fulfilling either of the following conditions:

i. With unsuccessful Kasai portoenterostomy procedure with a bilirubin >2 mg/dL, or ii. Who did not underwent Kasai portoenterostomy, or iii. With successful Kasai portoenterostomy procedure with a bilirubin <2 mg/dL, but with features of portal hypertension i.e. clinical splenomegaly and/or thrombocytopenia (platelets < 1,00,000/mm3).

Exclusion Criteria:

i. History suggestive of hyper-reactive airway disease. ii. Congestive heart failure iii. Any degree of heart block (I,, II, III) iv. Infants and children already on beta-blockers in last 4 weeks. v. Portal vein atresia or thrombosis. vi. History of variceal bleed. vii. Infants and children on prophylactic or therapeutic endotherapy (band ligation or sclerotherapy).

viii. Potential liver transplant within 1 month.

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 92 (Estimated)
Dates: Start 2020-08-15 (Actual); Primary Completion 2022-06-13 (Estimated); Study Completion 2022-06-15 (Estimated)

PRIMARY OUTCOMES:
Bleeding free survival over 18 months follow-up | 18 months

SECONDARY OUTCOMES:
Progression, persistence or regression of esophageal varices | 3 months
Progression, persistence or regression of gastric varices | 3 months
Progression, persistence or regression of portal hypertensive gastropathy | 3 months
Progression, persistence or regression of esophageal varices | 6 months
Progression, persistence or regression of gastric varices | 6 months
Progression, persistence or regression of portal hypertensive gastropathy | 6 months
Progression, persistence or regression of esophageal varices | 12 months
Progression, persistence or regression of gastric varices | 12 months
Progression, persistence or regression of portal hypertensive gastropathy | 12 months
Progression, persistence or regression of esophageal varices | 18 months
Progression, persistence or regression of gastric varices | 18 months
Progression, persistence or regression of portal hypertensive gastropathy | 18 months
Overall survival | 6 months
Overall survival | 12 months
Overall survival | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Rajeev Khanna, MD, Principal Investigator — Associate Professor, Pediatric Hepatology, Institute of Liver and Biliary Sciences
Locations (1):
- Institute of Liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided
Endoscopic details of the patients on propanolol or placebo

REFERENCES:
- [Background] Duche M, Ducot B, Ackermann O, Guerin F, Jacquemin E, Bernard O. Portal hypertension in children: High-risk varices, primary prophylaxis and consequences of bleeding. J Hepatol. 2017 Feb;66(2):320-327. doi: 10.1016/j.jhep.2016.09.006. Epub 2016 Sep 20. PMID 27663417
- [Background] Fagundes ED, Ferreira AR, Roquete ML, Penna FJ, Goulart EM, Figueiredo Filho PP, Bittencourt PF, Carvalho SD, Albuquerque W. Clinical and laboratory predictors of esophageal varices in children and adolescents with portal hypertension syndrome. J Pediatr Gastroenterol Nutr. 2008 Feb;46(2):178-83. doi: 10.1097/MPG.0b013e318156ff07. PMID 18223377
- [Background] Poddar U, Thapa BR, Rao KL, Singh K. Etiological spectrum of esophageal varices due to portal hypertension in Indian children: is it different from the West? J Gastroenterol Hepatol. 2008 Sep;23(9):1354-7. doi: 10.1111/j.1440-1746.2007.05102.x. Epub 2007 Aug 6. PMID 17683492
- [Background] Zargar SA, Javid G, Khan BA, Yattoo GN, Shah AH, Gulzar GM, Singh J, Rehman BU, Din Z. Endoscopic ligation compared with sclerotherapy for bleeding esophageal varices in children with extrahepatic portal venous obstruction. Hepatology. 2002 Sep;36(3):666-72. doi: 10.1053/jhep.2002.35278. PMID 12198659
- [Background] Zargar SA, Yattoo GN, Javid G, Khan BA, Shah AH, Shah NA, Gulzar GM, Singh J, Shafi HM. Fifteen-year follow up of endoscopic injection sclerotherapy in children with extrahepatic portal venous obstruction. J Gastroenterol Hepatol. 2004 Feb;19(2):139-45. doi: 10.1111/j.1440-1746.2004.03224.x. PMID 14731122
- [Background] Duche M, Ducot B, Tournay E, Fabre M, Cohen J, Jacquemin E, Bernard O. Prognostic value of endoscopy in children with biliary atresia at risk for early development of varices and bleeding. Gastroenterology. 2010 Dec;139(6):1952-60. doi: 10.1053/j.gastro.2010.07.004. Epub 2010 Jul 14. PMID 20637201
- [Background] Duche M, Ducot B, Ackermann O, Baujard C, Chevret L, Frank-Soltysiak M, Jacquemin E, Bernard O. Experience with endoscopic management of high-risk gastroesophageal varices, with and without bleeding, in children with biliary atresia. Gastroenterology. 2013 Oct;145(4):801-7. doi: 10.1053/j.gastro.2013.06.022. Epub 2013 Jun 19. PMID 23792202
- [Background] Shashidhar H, Langhans N, Grand RJ. Propranolol in prevention of portal hypertensive hemorrhage in children: a pilot study. J Pediatr Gastroenterol Nutr. 1999 Jul;29(1):12-7. doi: 10.1097/00005176-199907000-00007. PMID 10400097
- [Background] Drolet BA, Frommelt PC, Chamlin SL, Haggstrom A, Bauman NM, Chiu YE, Chun RH, Garzon MC, Holland KE, Liberman L, MacLellan-Tobert S, Mancini AJ, Metry D, Puttgen KB, Seefeldt M, Sidbury R, Ward KM, Blei F, Baselga E, Cassidy L, Darrow DH, Joachim S, Kwon EK, Martin K, Perkins J, Siegel DH, Boucek RJ, Frieden IJ. Initiation and use of propranolol for infantile hemangioma: report of a consensus conference. Pediatrics. 2013 Jan;131(1):128-40. doi: 10.1542/peds.2012-1691. Epub 2012 Dec 24. PMID 23266923